CLINICAL TRIAL: NCT03638011
Title: A Comparison of the Post-cesarean Section Analgesic Effects of Neuraxial Duramorph vs. Bilateral Transverse Abdominal Plane Block With Combined Bupivacaine/Liposomal Bupivacaine (Exparel)
Brief Title: A Comparison of the Post-C/S Analgesic Effects of Neuraxial Duramorph vs Bilateral TAP Block With Liposomal Bupivacaine
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Standard of Care changed due to COVID-19 and thus had to stop the study.
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, kalpana tyagaraj, Director of OB anesthesia, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-04-01-MMC
Record Dates: First submitted 2018-07-09; First posted 2018-08-20 (Actual); Results first posted 2021-03-03 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Caesarean Section
Keywords: Cesarean Section; Pregnancy

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized study evaluating the effectiveness of abdominal analgesia when using 266 mg EXPAREL delivered into the bilateral TAP blocks. TAP blocks are an excellent method for providing adequate analgesia following lower abdominal surgery.
  Those patients who wish to participate will be asked to sign a study consent form. Patients that decide to participate in this study will be randomized to either group 1 or group 2 (like the flip of a coin). Both groups will receive standard neuraxial anesthesia for their Cesarean Section and post-operative standard of care breakthrough medications for post-operative pain control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care (No Intervention): These participant will receive standard neuraxial anesthesia for their Cesarean Section and post-operative standard of care breakthrough medications for post-operative pain control. They standard neuraxial anesthesia with neuraxial Duramorph for post-operative pain.
- Bilateral TAP Block (Active Comparator): These participants will receive standard neuraxial anesthesia for their Cesarean Section and post-operative standard of care breakthrough medications for post-operative pain control. They will receive standard neuraxial anesthesia without neuraxial Duramorph and a transverse abdominal plane (TAP) blocks immediately after surgery, with a mixture of bupivacaine and Exparel, for post-operative analgesia.
  Interventions: Drug: Exparel

INTERVENTIONS:
Drug: Exparel — Bilateral TAP Blocks with combination of regular Bupivacaine and EXPAREL
  Other Names: TAP Block
  Arms: Bilateral TAP Block

SUMMARY:
The primary objective is to reduce or eliminate the use of all narcotics/opiates for post Cesarean section pain management. The investigators hypothesize that in comparison with epidural or intrathecal Duramorph, a TAP block with liposomal bupivacaine (Exparel) will provide better, longer-acting pain control and will significantly reduce the use of post-operative IV or p.o. opiates. This is a prospective, randomized clinical trial.

DETAILED DESCRIPTION:
The investigators will compare the analgesic efficacy and duration of an ultrasound guided bilateral TAP Block (with combined bupivacaine and liposomal bupivacaine) to Duramorph (an opiate). Neuraxial duramorph provides approximately 24 hours of pain relief (analgesia), whereas a bilateral TAP block with liposomal bupivacaine is expected to provide up to 72 hours of analgesia.

All participants will have neuraxial anesthesia (either a spinal or epidural) for their non-urgent or elective Cesarean section.

The control group (Group 1) will receive either intrathecal or epidural Duramorph (preservative-free morphine sulfate). Post-operatively, participants will have orders to receive, on an as-needed basis, IV/oral acetaminophen and/or IV/oral non-steroidal anti-inflammatory drugs (NSAIDS) for mild-moderate pain, and narcotics for severe pain; specifically- oxycodone or hydromorphone. All patients must receive acetaminophen and NSAIDS (unless contraindicated) before receiving narcotics. This multi-modal pain management regimen is our current standard of care.

The experimental group (Group 2) will also receive a spinal or epidural anesthetic. This group will not receive neuraxial Duramorph for post-operative pain. Instead, the patient will receive an ultrasound guided bilateral TAP block with a combination of bupivacaine and liposomal bupivacaine solution immediately after the Cesarean section. Additionally, all participants will receive the same post-operative analgesia orders as group 1.

ELIGIBILITY:
Inclusion Criteria:

* Females, aged 18-45 years inclusive and ASA physical status 1-3.
* Undergoing non-urgent Cesarean section with neuraxial anesthesia/analgesia.
* Subjects must be physically and mentally able to participate in the study and complete all study assessments.
* Subjects must be able to give fully informed consent to participate in this study after demonstrating a good understanding of the risks and benefits of the proposed components of the TAP infiltration.

Exclusion Criteria:

History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics

* Any subject whose anatomy, or surgical procedure, in the opinion of the Investigator, might preclude the potential successful performance of a bilateral TAP infiltration.
* Any subject who in the opinion of the Investigator, might be harmed or be a poor candidate for participation in the study.
* Any subject, who in the opinion of the Investigator, is on chronic pain medicine, including large doses of NSAIDs.
* Subjects who have received any investigational drug within 30 days prior to study drug administration, or planned administration of another investigational product or procedure during their participation in this study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — It is a status post C-section study.
Enrollment: 71 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kalpana Tyagaraj, MD, Principal Investigator — Maimonides Medical Center
Locations (2):
- United States (2):
  - Kalpana Tyagaraj, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bicket MC, Long JJ, Pronovost PJ, Alexander GC, Wu CL. Prescription Opioid Analgesics Commonly Unused After Surgery: A Systematic Review. JAMA Surg. 2017 Nov 1;152(11):1066-1071. doi: 10.1001/jamasurg.2017.0831. PMID 28768328
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Background] Johns N, O'Neill S, Ventham NT, Barron F, Brady RR, Daniel T. Clinical effectiveness of transversus abdominis plane (TAP) block in abdominal surgery: a systematic review and meta-analysis. Colorectal Dis. 2012 Oct;14(10):e635-42. doi: 10.1111/j.1463-1318.2012.03104.x. PMID 22632762
- [Background] Niraj G, Searle A, Mathews M, Misra V, Baban M, Kiani S, Wong M. Analgesic efficacy of ultrasound-guided transversus abdominis plane block in patients undergoing open appendicectomy. Br J Anaesth. 2009 Oct;103(4):601-5. doi: 10.1093/bja/aep175. Epub 2009 Jun 26. PMID 19561014
- [Background] Feierman DE, Kronenfeld M, Gupta PM, Younger N, Logvinskiy E. Liposomal bupivacaine infiltration into the transversus abdominis plane for postsurgical analgesia in open abdominal umbilical hernia repair: results from a cohort of 13 patients. J Pain Res. 2014 Aug 16;7:477-82. doi: 10.2147/JPR.S65151. eCollection 2014. PMID 25170277
- [Background] Dennis Feierman, Aden Bronstein, Miriam Flaum, Marc Dany Mohit Garg, Piyush Gupta and Kalpana Tyagaraj; A case series of 12 patient receiving bilateral Transverse Abdominis Plane blocks after cesarean section Open Journal of Anesthesiology December 2017: DOI: 10.4236/ ojanes.2017.712042
- [Background] Pack insert for Exparel

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Bilateral TAP Block
Started | 38 | 33
Completed | 38 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Bilateral TAP Block | Total
Number analyzed (Participants) | 38 | 33 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 33 | 71
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.08 (4.546) | 31.06 (4.062) | 31.07 (4.297)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 33 | 71
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 33 | 71

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessed by Visual Analog Scale (VAS) at 48 Hours
Description: To evaluate pain, participant will be shown a card that has a visual analogue (Faces) pains scale combined with numerical (0-10) analogue scale (0 is no pain, 10 is the worst pain imaginable).
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Bilateral TAP Block
Number analyzed (Participants) | 38 | 33
units on a scale | 1.97 (2.099) | 1.70 (2.084)

2. Primary Outcome: Pain Assessed by Visual Analog Scale (VAS) at 72 Hours
Description: as for outcome 1
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Bilateral TAP Block
Number analyzed (Participants) | 36 | 30
units on a scale | 0.67 (1.531) | 0.93 (1.574)

3. Secondary Outcome: Number of Participants Using Narcotics
Description: Total use of narcotics during the post operative period
Time Frame: 72 hours
Measure: Number; unit: participants
Arm/Group | Standard of Care | Bilateral TAP Block
Number analyzed (Participants) | 38 | 33
participants | 22 | 22

4. Secondary Outcome: Patient Satisfaction With Pain Control Assessed by 11 Point Satisfaction Scale
Description: Patient satisfaction with postsurgical pain management:
  0_____1_____2_____3_____4_____5_____6_____7_____8_____9_____10 0=not at all satisfied 10= extremely satisfied
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Bilateral TAP Block
Number analyzed (Participants) | 38 | 33
units on a scale | 9.18 (0.926) | 9.00 (1.904)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Standard of Care | Bilateral TAP Block
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/33
Other Adverse Events (participants affected / at risk) | 0/38 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT03638011/Prot_SAP_000.pdf